CLINICAL TRIAL: NCT06141044
Title: PANDREAS. Prophylactic Abdominal Drainage vs no Drainage After Distal Pancreatectomy: a Multicentre Clinical Trial
Brief Title: Prophylactic Abdominal Drainage vs no Drainage After Distal Pancreatectomy
Acronym: PANDREAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PANDREAS21101995
Record Dates: First submitted 2023-08-09; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pancreatic Fistula; Distal Pancreatectomy; Drainage
Keywords: Postoperative pancreatic fistula; Distal Pancreatectomy; Intraoperative Drainage

STUDY DESIGN:
Intervention Model Description: National, randomised, prospective, non-inferiority, multicentre clinical trial.To comparatively evaluate the rate of postoperative pancreatic fistula in patients undergoing distal pancreatectomy in one group with and one group without surgical drainage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drainage (No Intervention): Patients undergoing distal pancreatectomy with surgical drainage.
- No drainage (Experimental): Patients undergoing distal pancreatectomy without surgical drainage.
  Interventions: Procedure: Avoid surgical drainage

INTERVENTIONS:
Procedure: Avoid surgical drainage — Patients who undergo distal pancreatectomy, avoid placing a drain.
  Arms: No drainage

SUMMARY:
Postoperative pancreatic fistula (POPF) is a major source of morbidity and mortality after pancreatic resection, especially after distal pancreatectomy (PD). Today, POPF remains one of the main causes of hospital length of stay and healthcare costs. Numerous surgical techniques have been tested to reduce its incidence without success, so the current standard for the management of POPF, and the avoidance of associated complications, is intraoperative drain placement. However, surgically placed drains are not without risk. In recent years many studies, mostly retrospective, have attempted to determine whether omission of prophylactic drainage is associated with increased morbidity. These studies suggest that patients may benefit from not having a drain placed. This evidence challenges standard practice and the debate of whether or not to place a drain after distal pancreatectomy remains open. The investigators designed a prospective multicentre randomised non-inferiority study to determine whether prophylactic intraoperative drainage is associated with a lower morbidity rate after distal pancreatectomy.

DETAILED DESCRIPTION:
A prospective, randomised, multicentre, multicentre, randomised non-inferiority study is designed. The aim is to study whether patients who undergo distal pancreatectomy can benefit from the non-placement of a drain in terms of clinically relevant postoperative pancreatic fistula and Clavien-Dindo morbidity greater than or equal to 3.

Information will be collected for all patients undergoing distal pancreatectomy surgery at the collaborating centres who, upon invitation, voluntarily agree to participate in the study. Those who have agreed to participate, given written consent and meet the inclusion criteria and none of the exclusion criteria will be randomly assigned to one of the following treatment groups:

* Control group: patients who, after distal pancreatectomy, in whom abdominal drainage is placed.
* Intervention group: patients who, after distal pancreatectomy, will be omitted the placement of an abdominal drain.

Following the postoperative pancreatic fistula score according to the DISPAIR criteria, patients included in the present study will be stratified according to the preoperative risk of postoperative pancreatic fistula into: extreme, high, moderate and low.

The standards of surgical technique to be followed in both open and minimally invasive distal pancreatectomy were agreed by consensus.

Each patient will be followed up for 6 months from the time of randomisation (day of surgery).Those responsible for the recruitment and selection of patients for inclusion in the research project belong to the Multidisciplinary Committee of Hepatobiliary and Pancreatic Surgery of each centre. Surgical intervention, postoperative management and perioperative morbidity will be evaluated by the surgeon responsible for the patient. A patient recruitment period of 2 years is estimated. After a follow-up period of 6 months, an analysis of postoperative pancreatic fistula rate, perioperative morbidity, biochemical parameters and quality of life will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years of age) undergoing elective distal pancreatectomy surgery for any indication, with or without splenectomy, minimally invasive or open. It is not necessary to integrate gender perspective as it is not relevant and there is no influence on the results of POPF or morbidity.
* Signed informed consent was obtained from each of the patients included in the study.

Exclusion criteria

* Patients undergoing distal pancreatectomy as a secondary procedure
* Additional liver, gastric or colonic resection
* Pregnancy
* Participation in another study
* History of previous surgery involving the pancreas
* Patients with American Society of Anaesthesiologists classification 4
* Arterial resection other than the splenic artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant postoperative pancreatic fistula | From first postoperative day until day 30 after surgery
  The investigators define a clinically relevant pancreatic fistula following the 2016 update of the International Study Group (ISGPS) definition. According to this, a Clinically Relevant Postoperative Pancreatic Fistula refers to a grade B or C. Grade B requires a change in the postoperative management; drains are either left in place >3 weeks or repositioned through endoscopic or percutaneous procedures. Grade C postoperative pancreatic fistula refers to those postoperative pancreatic fistula that require reoperation or lead to single or multiple organ failure and/or mortality attributable to the pancreatic fistula.

SECONDARY OUTCOMES:
Clavien-Dindo morbidity greater than or equal to 3. | From first postoperative day until the ninth month after surgery
  To evaluate postoperative morbidity (Clavien-Dindo 3 or higher complications) in patients who undergo distal pancreatectomy. Comparing between the two groups of patients if there are any differences due to the presence or absence of a drainage.
  According to the Clavien-Dindo classification:
  3 - Requiring surgical, endoscopic or radiological intervention 3a-Intervention under regional/local anesthesia 3b- Intervention under general anesthesia 4 -Life-threatening complication requiring intensive care/intensive care unit management 4a- Single organ dysfunction 4b- Multi-organ dysfunction 5 - Patient demise
Reoperation. | From first postoperative day until day 90 after surgery
  To determine the rates of reoperation 90 days after distal pancreatectomy
Percutaneous drainage. | From first postoperative day until day 90 after surgery
  To determine the rates of percutaneous drainage 90 days after distal pancreatectomy. The need for a percutaneous drainage procedure, using an endoscopic or radiological approach, for the treatment of postoperative pancreatic fistula.
Abdominal collections | From first postoperative day until day 90 after surgery
  To determine the rate of abdominal collections 90 days after distal pancreatectomy. The investigators define an abdominal collection as a presence of liquid in the abdomen that cause symptoms in the patient, such as fever, and that may require less invasive therapeutic agents and treatment or percutaneous, endoscopic or angiographic interventional procedures.
Surgical wound infection. | From first postoperative day until day 90 after surgery
  To determine the rates of surgical site infection after distal pancreatectomy. Surgical site infection (SSI) is classified according to the Center for Disease Control and Prevention definition.
Delayed gastric emptying. | From first postoperative day until day 90 after surgery
  To determine rates of delayed gastric emptying after distal pancreatectomy. Delayed gastric emptying represents the inability to return to a standard diet by the end of the first postoperative week and includes prolonged nasogastric intubation of the patient. Three different grades (A, B, and C) are defined based on the impact on the clinical course and on postoperative management, according to the definition by the International Study Group of Pancreatic Surgery (ISGPS).
Postoperative bleeding. | From first postoperative day until day 90 after surgery
  According to the definition by the International Study Group of Pancreatic Surgery (ISGPS), postpancreatectomy bleeding is defined by 3 parameters: onset, location, and severity. The onset is either early (< or =24 hours after the end of the index operation) or late (>24 hours). The location is either intraluminal or extraluminal. The severity of bleeding may be either mild or severe.
  Three different grades of postpancreatectomy hemorrhage (grades A, B, and C) are defined according to the time of onset, site of bleeding, severity, and clinical impact.
Blood transfusion. | From first postoperative day until day 90 after surgery
  To determine rates of blood transfusion, measured in red blood cell concentrates after distal pancreatectomy.
Length of hospital stay | From first postoperative day until day 90 after surgery
  To determine rates of length of hospital stay after distal pancreatectomy. The length of hospital stay will be measured in days.
In-hospital mortality. | From first postoperative day after surgery.
  To determine rates of in-hospital mortality after distal pancreatectomy. The investigators will collet how many patients die during the hospitalization after surgery.
Intensive care admission. | From first postoperative day until day 90 after surgery
  To determine rates of intensive care admission 90 days after distal pancreatectomy. The investigators will measure how many patients need an intensive care admission and how long after surgery.
Mortality. | From first postoperative day until day 90 after surgery
  To determine rates of mortality 90 days after distal pancreatectomy
Readmission. | From first postoperative day until day 90 after surgery
  To determine rates of readmission 90 days after distal pancreatectomy. The investigators will collect how many patients, after surgery, needed for a readmission.
To study the role of serum amylase in the development of postoperative pancreatic fistula. | From first postoperative day until the fifth day after surgery
  The relevance of some biochemical markers that, in an early stage, can predict the development of postoperative pancreatic fistula has recently been highlighted.
  The serum amylase will be measured in U/L.
To study the role of amylase production in drainage in the development of postoperative pancreatic fistula. | From first postoperative day until the fifth day after surgery
  These data will be analysed on the first, third and fifth postoperative day. Amylase concentration in surgical drainage: The amylase concentration in surgical drainage will be measured on postoperative days 1, 3 and 5 to assess the early diagnostic ability of postoperative pancreatic fistula, of a concentration greater than 2000U/L.
  Drainage fluid amylase production, U/day (the product of the drainage fluid amylase value U/L and the amount of drainage, mL/day) will also be measured.
To study the role of biochemical parameters C-Reactive Protein in the development of postoperative pancreatic fistula. | From first postoperative day until the fifth day after surgery
  C-reactive protein concentration will be performed on postoperative days 1, 3 and 5 to assess the early diagnostic capability of POPF of a CRP concentration greater than 100 mg/L.
To study the role of Neutrophil-Lymphocyte Ratio (NLR) in the development of postoperative pancreatic fistula. | From first postoperative day until the fifth day after surgery
  The neutrophil/lymphocyte ratio has been published as a biochemical marker for the development of postoperative pancreatic fistula in duodenopancreatectomy.
  The investigators propose its analysis as a secondary objective, in order to determine its role as an early biochemical marker of fistula after distal pancreatectomy.
  Haemogram for calculation of serum leukocyte count will be performed on postoperative days 1, 3 and 5 to assess the early diagnostic capability of postoperative pancreatic fistula of a NLR greater than 8.5 mg/dl on these postoperative days.
To identify subgroups of patients according to their risk for postoperative pancreatic fistula | From first postoperative day until the fifth day after surgery
  In order to obtain the best evidence, it is proposed not only to analyse differences in morbidity, but also to stratify patients by risk of postoperative pancreatic fistula after distal pancreatectomy, as it is unclear whether omitting routine drainage in subgroups at high risk of postoperative pancreatic fistula could increase the risk of complications.To stratify patients according to the risk of postoperative pancreatic fistula, the DISPAIR score will be used which takes into account three variables: transection site (neck versus body/tail), pancreatic thickness at the transection site and diabetes. These variables have been previously studied as risk factors associated with postoperative pancreatic fistula.
To analyse the quality of life of patients undergoing distal pancreatectomy | From first postoperative day until the ninth month after surgery
  To analyse the quality of life of patients undergoing distal pancreatectomy. Variations in patients' quality of life will be measured using the official European Organization for Research and Treatment of Cancer (EORTC) questionnaires QLQ-C30 (generic quality of life questionnaire for cancer patients) and QLQ-PAN26 (specific quality of life questionnaire for pancreatic cancer patients). Although these questionnaires were developed for cancer patients and pancreatic cancer patients, they are widely used to assess postoperative quality of life after pancreatic surgery.
To examine the relevance of the neutrophil-lymphocyte ratio in the exclusion of postoperative pancreatic fistula after distal pancreatectomy. | From first postoperative day until the fifth day after surgery
  To examine the relevance of the neutrophil-lymphocyte ratio in the exclusion of postoperative pancreatic fistula after distal pancreatectomy.
To compare the quality of life of patients who undergo distal pancreatectomy according to the placement or non-placement of an intraoperative drain | From first postoperative day until the ninth month after surgery
  To compare the quality of life of patients who undergo distal pancreatectomy according to the placement or non-placement of an intraoperative drain.
  Variations in patients' quality of life will be measured using the official European Organization for Research and Treatment of Cancer (EORTC). Although this questionnaires were developed for cancer patients and pancreatic cancer patients, they are widely used to assess postoperative quality of life after pancreatic surgery.
To compare the quality of life of patients who undergo distal pancreatectomy according to the placement or non-placement of an intraoperative drain | From first postoperative day until ninth month after surgery
  Variations in patients' quality of life will be measured using the QLQ-C30 (generic quality of life questionnaire for cancer patients).Although this questionnaires were developed for cancer patients and pancreatic cancer patients, they are widely used to assess postoperative quality of life after pancreatic surgery.
To compare the quality of life of patients who undergo distal pancreatectomy according to the placement or non-placement of an intraoperative drain | From first postoperative day until ninth month after surgery
  Variations in patients' quality of life will be measured using the QLQ-PAN26 (specific quality of life questionnaire for pancreatic cancer patients).Although this questionnaires were developed for cancer patients and pancreatic cancer patients, they are widely used to assess postoperative quality of life after pancreatic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rotellar, MD, PhD, Study Director — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
Databases with anonymized IPD will be shared at the end of the study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available at the completion of the study and will remain available from that moment onward.
Access Criteria: Upon request to researchers

REFERENCES:
- [Background] Lillemoe KD, Kaushal S, Cameron JL, Sohn TA, Pitt HA, Yeo CJ. Distal pancreatectomy: indications and outcomes in 235 patients. Ann Surg. 1999 May;229(5):693-8; discussion 698-700. doi: 10.1097/00000658-199905000-00012. PMID 10235528
- [Background] Balcom JH 4th, Rattner DW, Warshaw AL, Chang Y, Fernandez-del Castillo C. Ten-year experience with 733 pancreatic resections: changing indications, older patients, and decreasing length of hospitalization. Arch Surg. 2001 Apr;136(4):391-8. doi: 10.1001/archsurg.136.4.391. PMID 11296108
- [Background] Kleeff J, Diener MK, Z'graggen K, Hinz U, Wagner M, Bachmann J, Zehetner J, Muller MW, Friess H, Buchler MW. Distal pancreatectomy: risk factors for surgical failure in 302 consecutive cases. Ann Surg. 2007 Apr;245(4):573-82. doi: 10.1097/01.sla.0000251438.43135.fb. PMID 17414606
- [Background] Sledzianowski JF, Duffas JP, Muscari F, Suc B, Fourtanier F. Risk factors for mortality and intra-abdominal morbidity after distal pancreatectomy. Surgery. 2005 Feb;137(2):180-5. doi: 10.1016/j.surg.2004.06.063. PMID 15674199
- [Background] Nathan H, Cameron JL, Goodwin CR, Seth AK, Edil BH, Wolfgang CL, Pawlik TM, Schulick RD, Choti MA. Risk factors for pancreatic leak after distal pancreatectomy. Ann Surg. 2009 Aug;250(2):277-81. doi: 10.1097/SLA.0b013e3181ae34be. PMID 19638926
- [Background] Pannegeon V, Pessaux P, Sauvanet A, Vullierme MP, Kianmanesh R, Belghiti J. Pancreatic fistula after distal pancreatectomy: predictive risk factors and value of conservative treatment. Arch Surg. 2006 Nov;141(11):1071-6; discussion 1076. doi: 10.1001/archsurg.141.11.1071. PMID 17116799
- [Background] Knaebel HP, Diener MK, Wente MN, Buchler MW, Seiler CM. Systematic review and meta-analysis of technique for closure of the pancreatic remnant after distal pancreatectomy. Br J Surg. 2005 May;92(5):539-46. doi: 10.1002/bjs.5000. PMID 15852419
- [Background] Karabicak I, Satoi S, Yanagimoto H, Yamamoto T, Yamaki S, Kosaka H, Hirooka S, Kotsuka M, Michiura T, Inoue K, Matsui Y, Kon M. Comparison of surgical outcomes of three different stump closure techniques during distal pancreatectomy. Pancreatology. 2017 May-Jun;17(3):497-503. doi: 10.1016/j.pan.2017.04.005. Epub 2017 Apr 8. PMID 28411019
- [Background] Ecker BL, McMillan MT, Allegrini V, Bassi C, Beane JD, Beckman RM, Behrman SW, Dickson EJ, Callery MP, Christein JD, Drebin JA, Hollis RH, House MG, Jamieson NB, Javed AA, Kent TS, Kluger MD, Kowalsky SJ, Maggino L, Malleo G, Valero V 3rd, Velu LKP, Watkins AA, Wolfgang CL, Zureikat AH, Vollmer CM Jr. Risk Factors and Mitigation Strategies for Pancreatic Fistula After Distal Pancreatectomy: Analysis of 2026 Resections From the International, Multi-institutional Distal Pancreatectomy Study Group. Ann Surg. 2019 Jan;269(1):143-149. doi: 10.1097/SLA.0000000000002491. PMID 28857813
- [Background] Bassi C, Molinari E, Malleo G, Crippa S, Butturini G, Salvia R, Talamini G, Pederzoli P. Early versus late drain removal after standard pancreatic resections: results of a prospective randomized trial. Ann Surg. 2010 Aug;252(2):207-14. doi: 10.1097/SLA.0b013e3181e61e88. PMID 20622661
- [Background] Conlon KC, Labow D, Leung D, Smith A, Jarnagin W, Coit DG, Merchant N, Brennan MF. Prospective randomized clinical trial of the value of intraperitoneal drainage after pancreatic resection. Ann Surg. 2001 Oct;234(4):487-93; discussion 493-4. doi: 10.1097/00000658-200110000-00008. PMID 11573042
- [Background] Mangieri CW, Kuncewitch M, Fowler B, Erali RA, Moaven O, Shen P, Clark CJ. Surgical drain placement in distal pancreatectomy is associated with an increased incidence of postoperative pancreatic fistula and higher readmission rates. J Surg Oncol. 2020 Sep;122(4):723-728. doi: 10.1002/jso.26072. Epub 2020 Jul 2. PMID 32614999
- [Background] Paulus EM, Zarzaur BL, Behrman SW. Routine peritoneal drainage of the surgical bed after elective distal pancreatectomy: is it necessary? Am J Surg. 2012 Oct;204(4):422-7. doi: 10.1016/j.amjsurg.2012.02.005. Epub 2012 May 10. PMID 22579230
- [Background] Behrman SW, Zarzaur BL, Parmar A, Riall TS, Hall BL, Pitt HA. Routine drainage of the operative bed following elective distal pancreatectomy does not reduce the occurrence of complications. J Gastrointest Surg. 2015 Jan;19(1):72-9; discussion 79. doi: 10.1007/s11605-014-2608-z. Epub 2014 Aug 13. PMID 25115324
- [Background] Correa-Gallego C, Brennan MF, D'angelica M, Fong Y, Dematteo RP, Kingham TP, Jarnagin WR, Allen PJ. Operative drainage following pancreatic resection: analysis of 1122 patients resected over 5 years at a single institution. Ann Surg. 2013 Dec;258(6):1051-8. doi: 10.1097/SLA.0b013e3182813806. PMID 23360918
- [Background] Vissers FL, Balduzzi A, van Bodegraven EA, van Hilst J, Festen S, Hilal MA, Asbun HJ, Mieog JSD, Koerkamp BG, Busch OR, Daams F, Luyer M, De Pastena M, Malleo G, Marchegiani G, Klaase J, Molenaar IQ, Salvia R, van Santvoort HC, Stommel M, Lips D, Coolsen M, Bassi C, van Eijck C, Besselink MG; Dutch Pancreatic Cancer Group. Prophylactic abdominal drainage or no drainage after distal pancreatectomy (PANDORINA): a binational multicenter randomized controlled trial. Trials. 2022 Sep 24;23(1):809. doi: 10.1186/s13063-022-06736-5. PMID 36153559
- [Background] Van Buren G 2nd, Bloomston M, Schmidt CR, Behrman SW, Zyromski NJ, Ball CG, Morgan KA, Hughes SJ, Karanicolas PJ, Allendorf JD, Vollmer CM Jr, Ly Q, Brown KM, Velanovich V, Winter JM, McElhany AL, Muscarella P 2nd, Schmidt CM, House MG, Dixon E, Dillhoff ME, Trevino JG, Hallet J, Coburn NSG, Nakeeb A, Behrns KE, Sasson AR, Ceppa EP, Abdel-Misih SRZ, Riall TS, Silberfein EJ, Ellison EC, Adams DB, Hsu C, Tran Cao HS, Mohammed S, Villafane-Ferriol N, Barakat O, Massarweh NN, Chai C, Mendez-Reyes JE, Fang A, Jo E, Mo Q, Fisher WE. A Prospective Randomized Multicenter Trial of Distal Pancreatectomy With and Without Routine Intraperitoneal Drainage. Ann Surg. 2017 Sep;266(3):421-431. doi: 10.1097/SLA.0000000000002375. PMID 28692468
- [Background] van Bodegraven EA, van Ramshorst TME, Balduzzi A, Hilal MA, Molenaar IQ, Salvia R, van Eijck C, Besselink MG. Routine abdominal drainage after distal pancreatectomy: meta-analysis. Br J Surg. 2022 May 16;109(6):486-488. doi: 10.1093/bjs/znac042. No abstract available. PMID 35576374
- [Background] van Bodegraven EA, De Pastena M, Vissers FL, Balduzzi A, Stauffer J, Esposito A, Malleo G, Marchegiani G, Busch OR, Salvia R, van Hilst J, Bassi C, Besselink MG, Asbun HJ. Routine prophylactic abdominal drainage versus no-drain strategy after distal pancreatectomy: A multicenter propensity score matched analysis. Pancreatology. 2022 Sep;22(6):797-802. doi: 10.1016/j.pan.2022.06.002. Epub 2022 Jun 2. PMID 35690539
- [Background] Bonsdorff A, Ghorbani P, Helantera I, Tarvainen T, Kontio T, Belfrage H, Siren J, Kokkola A, Sparrelid E, Sallinen V. Development and external validation of DISPAIR fistula risk score for clinically relevant postoperative pancreatic fistula risk after distal pancreatectomy. Br J Surg. 2022 Oct 14;109(11):1131-1139. doi: 10.1093/bjs/znac266. PMID 35983583
- [Background] Hirono S, Kawai M, Okada KI, Miyazawa M, Kitahata Y, Kobayashi R, Hayata K, Hayami S, Ueno M, Yamaue H. Division of the pancreas at the neck reduces postoperative pancreatic fistula in laparoscopic distal pancreatectomy: Comparison of pancreatic division at the body. Pancreatology. 2021 Mar;21(2):480-486. doi: 10.1016/j.pan.2020.12.021. Epub 2021 Jan 4. PMID 33518455
- [Background] Asbun HJ, Van Hilst J, Tsamalaidze L, Kawaguchi Y, Sanford D, Pereira L, Besselink MG, Stauffer JA. Technique and audited outcomes of laparoscopic distal pancreatectomy combining the clockwise approach, progressive stepwise compression technique, and staple line reinforcement. Surg Endosc. 2020 Jan;34(1):231-239. doi: 10.1007/s00464-019-06757-3. Epub 2019 May 28. PMID 31139993
- [Background] Sell NM, Pucci MJ, Gabale S, Leiby BE, Rosato EL, Winter JM, Yeo CJ, Lavu H. The influence of transection site on the development of pancreatic fistula in patients undergoing distal pancreatectomy: A review of 294 consecutive cases. Surgery. 2015 Jun;157(6):1080-7. doi: 10.1016/j.surg.2015.01.014. Epub 2015 Mar 16. PMID 25791028
- [Background] Pecorelli N, Guarneri G, Palucci M, Gozzini L, Vallorani A, Crippa S, Partelli S, Falconi M. Early biochemical predictors of clinically relevant pancreatic fistula after distal pancreatectomy: a role for serum amylase and C-reactive protein. Surg Endosc. 2022 Jul;36(7):5431-5441. doi: 10.1007/s00464-021-08883-3. Epub 2022 Jan 6. PMID 34988737
- [Background] Sakamoto K, Ogawa K, Tamura K, Iwata M, Matsui T, Nishi Y, Nagaoka T, Funamizu N, Takai A, Takada Y. Postoperative elevation of C-reactive protein levels and high drain fluid amylase output are strong predictors of pancreatic fistulas after distal pancreatectomy. J Hepatobiliary Pancreat Sci. 2021 Oct;28(10):874-882. doi: 10.1002/jhbp.927. Epub 2021 Mar 16. PMID 33636044
- [Background] Garnier J, Alfano MS, Robin F, Ewald J, Al Farai A, Palen A, Sebai A, Mokart D, Delpero JR, Sulpice L, Zemmour C, Turrini O. Establishment and external validation of neutrophil-to-lymphocyte ratio in excluding postoperative pancreatic fistula after pancreatoduodenectomy. BJS Open. 2023 Jan 6;7(1):zrac124. doi: 10.1093/bjsopen/zrac124. PMID 36633417
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957